CLINICAL TRIAL: NCT03155243
Title: Impact of Humira® Therapy on Ocular Inflammation, Selected Health Care Resource Utilization and Patient Reported Outcomes in Patients With Active Non-infectious Intermediate, Posterior and Panuveitis in Routine Clinical Practice -HOPE
Brief Title: Impact of Humira® Therapy on Ocular Inflammation, Selected Health Care Resource Utilization and Patient Reported Outcomes in Patients With Active Non-infectious Intermediate, Posterior and Panuveitis in Routine Clinical Practice
Acronym: HOPE
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P16-537
Record Dates: First submitted 2017-05-15; First posted 2017-05-16 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Uveitis
Keywords: Humira®; Adalimumab; Ocular inflammation; Active non-infectious intermediate, posterior and panuveitis
MeSH Terms: conditions — Uveitis; Panuveitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants receiving adalimumab (Humira®): Participants with active non- infectious intermediate, posterior or panuveitis receiving adalimumab (Humira®).

SUMMARY:
This study aims at evaluating real life effectiveness of originator adalimumab (Humira®) participants with active non-infectious intermediate, posterior and panuveitis (NIIPPU) despite high-dose corticosteroid therapy; including effect on ocular inflammation, health-related quality of life, health resource utilization, work ability and medication burden, as well as describe the characteristics of NIIPPU participants treated with Humira® in the real-life setting.

ELIGIBILITY:
Inclusion Criteria:

* Participants voluntarily signed a patient authorization form to use and disclose personal health information (or informed consent, where applicable).
* Age >= 18 years at the time of the enrollment.
* Diagnosis of active NIIPP uveitis as defined by the presence of at least 1 of the following parameters:

  1. Active, inflammatory, chorioretinal and/or inflammatory retinal vascular lesion
  2. >= 2+ anterior chamber cells [Standardization of Uveitis Nomenclature (SUN) criteria]
  3. >= 2+ vitreous haze [National Eye Institute (NEI)/SUN criteria]
* Humira® treatment is indicated as per local Summary of Product Characteristics (SmPC) and professional and/or reimbursement guidelines.
* Decision on the treatment with Humira® was made prior to any decision to approach the patient to participate in this study.

Exclusion Criteria:

* Participants who cannot be treated with Humira® according to the local Humira® SmPC and/or local professional and reimbursement guidelines.
* Prior treatment with Humira®, including current course of Humira® started prior to baseline visit assessments.
* Participants currently participating in other clinical research.
* Participants who are unwilling or unable to complete the quality of life and other patient reported questionnaires.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with diagnosed active non- infectious intermediate, posterior or panuveitis (NIIPPU) that are being treated with Humira® as per locally approved label and prescription guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who achieve treatment response at any of the follow-up visits | Up to Month 12
  Definition of response: "quiescence" defined as patients with no new active chorioretinal inflammatory lesions and having anterior chamber (AC) cell and vitreous haze (VH) grade of <=0.5+ in both eyes.

SECONDARY OUTCOMES:
Proportion of participants with maintained response at any of follow up visits | Up to Month 12
  Maintained response is defined as quiescence achieved at respective prior visit and no flare at current visit.
Percent change in Presenteeism | Up to Month 12
  Assessing percent change in presenteeism
Proportion of participants with maintained response separately for each follow-up visit | Up to Month 12
  Maintained response is defined as quiescence achieved at respective prior visit and no flare at current visit.
Percent Change in Total activity impairment | Up to Month 12
  Assessing Percent Change in Total activity impairment
Changes in total score of Work Productivity & Activity Impairment (WPAI)-UV score | From Month 1 to Month 12
  Assessing changes in total score of WPAI-UV score
Change in emergency room admissions | From 6 months prior to treatment start (Week 0 [baseline]) to 12 months after treatment start (total 18 months)
  Assessing change in emergency room admissions
Proportion of participants with treatment response separately for each follow-up visit | Up to Month 12
  Response is defined as participants with no new active inflammatory lesions and having anterior chamber (AC) cell and vitreous haze (VH) grade of <=0.5+ in both eyes.
Change from baseline in Best corrected visual acuity (BCVA) | From Month 1 to Month 12
  Assessing change from baseline in Best corrected visual acuity (BCVA)
Change in cumulative hospital admissions | From 6 months prior to treatment start (Week 0 [baseline]) to 12 months after treatment start (total 18 months)
  Assessing change in cumulative hospital admissions
Change from baseline in Central Retinal Thickness (CRT) | From 6 months prior to treatment start (Week 0 [baseline]) to 12 months after treatment start (total 18 months)
  Assessing change from baseline in Central Retinal Thickness (CRT)
Proportion of participants with flare at any of follow up visit | Up to Month 12
  Flare is defined as new active inflammatory lesions or AC cell grade of >=2+ or VH grade of >=2+ at least in one eye.
Percent change in Absenteeism | Up to Month 12
  Assessing percent change in absenteeism
Percent Change in Total work productivity impairment | Up to Month 12
  Assessing Percent Change in Total work productivity impairment
Change in outpatient visits | From 6 months prior to treatment start (Week 0 [baseline]) to 12 months after treatment start (total 18 months)
  Assessing change in outpatient visits
Change in hospitalization days prior to and during Humira® treatment | From 6 months prior to treatment start (Week 0 [baseline]) to 12 months after treatment start (total 18 months)
  Assessing change in hospitalization days prior to and during Humira® treatment
Change from baseline in intraocular pressure | From Month 1 to Month 12
  Assessing change from baseline in intraocular pressure

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (28):
- Austria (2):
  - Medizinische Universität Graz /ID# 206301, Graz, Styria
  - Medical University of Vienna /ID# 206190, Vienna, Vienna
- Colombia (3):
  - Clinica Oftalmologica del Caribe /ID# 206448, Barranquilla, Atlántico
  - Foscal /Id# 207362, Bucaramanga
  - Fundacion hospitalaria San Vicente de Paul /ID# 208295, Medellín
- Vseobecna Fakultni Nemocnice /ID# 209530, Prague, Czechia
- Germany (3):
  - Charite Campus Virchow-Klinikum /ID# 204879, Berlin
  - Universitätsklinikum Hamburg-Eppendorf /ID# 205234, Hamburg
  - St. Franziskus Hosp Muenster /ID# 206695, Münster
- Greece (4):
  - Omma /Id# 163750, Athens
  - Athens Eye Hospital /ID# 163751, Athens
  - University General Hospital of Ioannina /ID# 163752, Ioannina
  - Interbalkan Medical Center /ID# 163753, Thessaloniki
- Hungary (2):
  - Semmelweis Egyetem /ID# 163647, Budapest
  - Szegedi Tudomanyegyetem /ID# 163646, Szeged
- Royal Victoria Eye and Ear Hos /ID# 163653, Dublin, Ireland
- Israel (6):
  - Hadassah Medical Center /ID# 169305, Jerusalem, Jerusalem
  - Rabin Medical Center /ID# 163108, Petakh Tikva, Tel Aviv
  - Tel Aviv Sourasky Medical Ctr /ID# 163024, Tel Aviv, Tel Aviv
  - Barzilai Medical Center /ID# 163025, Ashkelon
  - Bnai Zion Medical Center /ID# 163026, Haifa
  - Sheba Medical Center /ID# 163109, Ramat Gan
- Albahar Ophtalmology Center /ID# 210124, Kuwait City, Kuwait
- American University of Beirut /ID# 210122, Beirut, Lebanon
- Switzerland (3):
  - Stadtspital Triemli /ID# 206204, Zurich, Canton of Zurich
  - Inselspital, Universitaetsklinik /ID# 201027, Bern
  - Hop Ophtalmique Jules Gonin /ID# 201028, Lausanne
- Cleveland Clinic Abu Dhabi /ID# 210123, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvie.com/content/dam/abbvie-dotcom/clinical-trials/adalimumab_P16-537.pdf